CLINICAL TRIAL: NCT07190248
Title: A Phase 3, Randomized, Open-label, Multicenter Clinical Study to Evaluate the Safety and Efficacy of MK-1084 in Combination With Subcutaneous Pembrolizumab and Berahyaluronidase Alfa (MK-3475A) Versus MK-3475A in Combination With Pemetrexed/Platinum (Carboplatin or Cisplatin) Chemotherapy as First-line Treatment of Participants With KRAS G12C-Mutant, Advanced or Metastatic Nonsquamous NSCLC (KANDLELIT-007)
Brief Title: A Clinical Study of Calderasib (MK-1084) and Other Treatments for Participants With Non-Small Cell Lung Cancer (MK-1084-007/KANDLELIT-007)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1084-007; U1111-1307-9569 (Registry Identifier: UTN); 2024-514500-14-00 (Registry Identifier: EU CT); MK-1084-007 (Other: MSD); KANDLELIT-007 (Other: MSD); jRCT2031240722 (Registry Identifier: Registry Identifier Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Calderasib + Pembrolizumab (+) Berahyaluronidase alfa (Experimental): Participants will receive pembrolizumab (+) berahyaluronidase alfa at a fixed dose subcutaneously on Day 1 of each 6-week cycle for up to 18 cycles (approximately 2 years) plus calderasib until discontinuation criterion is met.
  Interventions: Drug: Calderasib; Biological: Pembrolizumab (+) Berahyaluronidase alfa
- Pembrolizumab (+) Berahyaluronidase alfa + Chemotherapy (Active Comparator): Participants will receive pembrolizumab (+) berahyaluronidase alfa at a fixed dose subcutaneously on Day 1 of each 6-week cycle for up to 18 cycles (approximately 2 years) and pemetrexed via intravenous (IV) infusion at a dose of 500 mg/m^2 on days 1 and 22 of cycles 1 and 3 until discontinuation criterion is met PLUS investigator's choice of carboplatin via IV infusion at area under curve (AUC) 5 mg/mL/minute on days 1 and 22 of cycles 1 and 3 (up to 4 doses, approximately 6 weeks) OR cisplatin via IV infusion at a dose of 75 mg/m^2 on days 1 and 22 of cycles 1 and 3 (up to 4 doses, approximately 6 weeks).
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Calderasib — Administered as an oral tablet
  Other Names: MK-1084
  Arms: Calderasib + Pembrolizumab (+) Berahyaluronidase alfa
Biological: Pembrolizumab (+) Berahyaluronidase alfa — Administered as a SC injection
  Other Names: MK-3475A
Drug: Pemetrexed — Administered as an IV Infusion
  Other Names: Alimta
  Arms: Pembrolizumab (+) Berahyaluronidase alfa + Chemotherapy
Drug: Cisplatin — Administered as an IV Infusion
  Other Names: Platinol-AQ
  Arms: Pembrolizumab (+) Berahyaluronidase alfa + Chemotherapy
Drug: Carboplatin — Administered as an IV Infusion
  Other Names: PARAPLATIN®
  Arms: Pembrolizumab (+) Berahyaluronidase alfa + Chemotherapy

SUMMARY:
Researchers want to learn if the study medicines calderasib and subcutaneous (SC) pembrolizumab can be used to treat non-small cell lung cancer (NSCLC) when given together. Calderasib is a targeted therapy for the KRAS G12C mutation.

The goal of this study is to learn if people who receive calderasib with SC pembrolizumab live longer without the cancer growing or spreading than in people who receive SC pembrolizumab with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has nonsquamous NSCLC (Stage IIIB, Stage IIIC) not eligible for curative resection or chemoradiation or Stage IV: M1a, M1b, or M1c
* If human immunodeficiency virus (HIV) positive, must have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous clear history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has a gastrointestinal disorder affecting absorption
* Is HIV positive and has a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has received prior systemic anticancer therapy for their advanced or metastatic NSCLC
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy except those specified by protocol
* Has history of stem cell/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2029-12-07 (Estimated); Study Completion 2032-08-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in Participants with Programmed Death-Ligand 1 (PD-L1) Tumor Proportion Score (TPS) ≥1% | Up to approximately 48 months
  PFS is defined as the time from randomization until either documented disease progression per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or death due to any cause, whichever occurs first. PFS as determined by blinded independent central review (BICR) will be presented.

SECONDARY OUTCOMES:
PFS in All Participants | Up to approximately 48 months
  PFS is defined as the time from randomization until either documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first. PFS as determined by BICR will be presented.
Overall Survival (OS) in Participants with PD-L1 TPS ≥1% | Up to approximately 62 months
  OS is defined as the time from randomization to death due to any cause.
OS in Participants in All Participants | Up to approximately 62 months
  OS is defined as the time from randomization to death due to any cause.
Overall Response Rate (ORR) in All Participants | Up to approximately 48 months
  ORR is defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) per RECIST1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.
ORR in Participants with PD-L1 TPS ≥1% | Up to approximately 48 months
  ORR is defined as the percentage of participants with CR or PR per RECIST1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Duration of Response (DOR) | Up to approximately 48 months
  For participants who demonstrate confirmed CR or PR per RECIST 1.1 as assessed by BICR, duration of response is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experienced One or More Adverse Events (AEs) | Up to approximately 81 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 81 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who discontinue study treatment due to an AE will be presented.
Change from Baseline in Global Health Status/Quality of Life (GHS/QoL) (Items 29, 30) on the European Organization for Research and Treatment of Cancer QoL Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline and up to approximately 81 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the score of EORTC QLQ-C30 Items 29 and 30 will be presented. Higher scores indicate a better overall health status.
Change from Baseline in Dyspnea Score (Item 8) on the EORTC QLQ-C30 | Baseline and up to approximately 81 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C30 Item 8 will be presented. A higher score indicates a worse level of dyspnea.
Change from Baseline in Cough Score (Item 31) on the European Organization for Research and Treatment of Cancer Quality of Life Lung Cancer-Specific Questionnaire (EORTC QLQ-LC13) | Baseline and up to approximately 81 months
  The EORTC QLQ-C13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C13 Item 31 will be presented. A higher score indicates more frequent coughing.
Change from Baseline in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 | Baseline and up to approximately 81 months
  The EORTC QLQ-C13 is lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C13 Item 40 will be presented. A higher score indicates a worse level of chest pain.
Time to Deterioration (TTD) in GHS/QoL (Items 29, 30) on the EORTC QLQ-C30 | Baseline and up to approximately 81 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in global health status (GHS) and quality of life (QoL) (EORTC QLQ-C30 Items 29 and 30) score. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in GHS and QoL, will be presented. A longer TTD indicates a better outcome.
TTD in Dyspnea Score (Item 8) on the EORTC QLQ-C30 | Baseline and up to approximately 81 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in dyspnea (EORTC QLQ-C30 Item 8) score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in dyspnea score, will be presented. A longer TTD indicates a better outcome.
TTD in Cough Score (Item 31) on the EORTC QLQ-LC13 | Baseline and up to approximately 81 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in cough (EORTC QLQ-C13 Item 31) score. The EORTC QLQ-C13 is lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in cough score, will be presented. A longer TTD indicates a better outcome.
TTD in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 | Baseline and up to approximately 81 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in chest pain (EORTC QLQ-C13 Item 40) score. The EORTC QLQ-C13 is lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline chest pain score, will be presented. A longer TTD indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (74):
- United States (7):
  - Central Alabama Research ( Site 0108), Birmingham, Alabama
  - Stamford Hospital ( Site 0126), Stamford, Connecticut
  - Mount Sinai Cancer Center ( Site 0137), Miami Beach, Florida
  - New England Cancer Specialists ( Site 0139), Westbrook, Maine
  - New York Oncology Hematology, P.C. ( Site 0119), Albany, New York
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute ( Site 0111), Lancaster, Pennsylvania
  - Blue Ridge Cancer Care ( Site 0144), Roanoke, Virginia
- Argentina (4):
  - Instituto Alexander Fleming ( Site 0311), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0300), Mar del Plata, Buenos Aires
  - Hospital Italiano de Cordoba ( Site 0308), Córdoba
  - CEMAIC ( Site 0309), Córdoba
- Australia (2):
  - Northern Beaches Hospital ( Site 2905), Frenchs Forest, New South Wales
  - Mater Hospital Brisbane ( Site 2906), South Brisbane, Queensland
- Medizinische Universität Graz-Klinische Abteilung für Pulmonologie ( Site 1005), Graz, Styria, Austria
- China (5):
  - Anhui Provincial Cancer Hospital ( Site 2708), Hefei, Anhui
  - Beijing Cancer hospital-Thoracic Cancer Department A ( Site 2700), Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University ( Site 2744), Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University ( Site 2704), Nanning, Guangxi
  - Sichuan Cancer Hospital. ( Site 2739), Chengdu, Sichuan
- France (7):
  - Hopital Europeen Marseille ( Site 1207), Marseille, Bouches-du-Rhone
  - CHU Caen ( Site 1212), Caen, Calvados
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois ( Site 1209), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Metropole Savoie Site de Chambery ( Site 1208), Chambéry, Savoie
  - Clinique de l'Europe ( Site 1213), Amiens, Somme
  - Groupe Hospitalier Paris Saint Joseph ( Site 1215), Paris
  - Hôpital Européen Georges Pompidou ( Site 1214), Paris
- Greece (4):
  - Agios Andreas Hospital Patras ( Site 1407), Pátrai, Achaia
  - Errikos Dunant Hospital Center ( Site 1408), Athens, Attica
  - Metropolitan General Hospital ( Site 1400), Athens, Attica
  - Papageorgiou General Hospital of Thessaloniki ( Site 1403), Thessaloniki
- Reformatus Pulmonologiai Centrum ( Site 1503), Törökbálint, Pest County, Hungary
- Israel (5):
  - Yitzhak Shamir Medical Center. ( Site 1709), Beer Ya Akov
  - Shaare Zedek Medical Center ( Site 1706), Jerusalem
  - Meir Medical Center. ( Site 1702), Kfar Saba
  - Sheba Medical Center ( Site 1700), Ramat Gan
  - Sourasky Medical Center ( Site 1705), Tel Aviv
- Italy (2):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII ( Site 1811), Bergamo, Lombardy
  - AOU Renato Dulbecco ( Site 1804), Catanzaro
- Japan (9):
  - National Hospital Organization Himeji Medical Center ( Site 2827), Himeji, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 2811), Kobe, Hyōgo
  - Matsusaka Municipal Hospital ( Site 2808), Matsusaka, Mie-ken
  - Tohoku University Hospital ( Site 2804), Sendai, Miyagi
  - Osaka Medical and Pharmaceutical University Hospital ( Site 2810), Takatsuki, Osaka
  - National Hospital Organization Ureshino Medical Center ( Site 2817), Ureshino, Saga-ken
  - Nippon Medical School Hospital ( Site 2819), Bunkyo, Tokyo
  - Tokyo Medical University Hospital ( Site 2829), Shinjuku, Tokyo
  - Osaka Metropolitan University Hospital ( Site 2826), Osaka
- Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 2012), Gliwice, Silesian Voivodeship, Poland
- Romania (5):
  - Institutul Oncologic Prof. Dr. I Chiricuta ( Site 2103), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL-Oncologie Medicala ( Site 2101), Florești, Cluj
  - SC ONCO CARD SRL ( Site 2109), Brasov
  - Delta Health Care SRL ( Site 2108), Bucharest
  - SC MNT Healthcare Europe SRL ( Site 2105), Bucharest
- South Korea (6):
  - Chonnam National University Hwasun Hospital ( Site 3502), Jeollanam-do, Jeonranamdo
  - Pusan National University Yangsan Hospital ( Site 3504), Yangsan, Kyongsangnam-do
  - Pusan National University Hospital ( Site 3501), Busan, Pusan-Kwangyokshi
  - Chungnam National University Hospital ( Site 3503), Daejeon, Taejon-Kwangyokshi
  - Kyung Hee University Medical Center ( Site 3500), Seoul
  - Korea University Guro Hospital ( Site 3505), Seoul
- Spain (6):
  - Institut Català d'Oncologia (ICO) - Badalona ( Site 2200), Badalona, Catalonia
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 2201), Barcelona, Catalonia
  - Complejo Hospitalario Universitario A Coruna ( Site 2207), A Coruña, La Coruna
  - Hospital General Universitario de Valencia ( Site 2204), Valencia, Valenciana, Comunitat
  - Hospital Universitario Ramon y Cajal ( Site 2203), Madrid
  - Hospital Universitario Virgen de Valme ( Site 2205), Seville
- Taiwan (5):
  - Chang Gung Memorial Hospital- Chiayi ( Site 3611), Chiayi City, Chiayi
  - Taipei Medical University Shuang Ho Hospital ( Site 3602), New Taipei City
  - National Cheng Kung University Hospital ( Site 3604), Tainan
  - MacKay Memorial Hospital ( Site 3609), Taipei
  - Tri-Service General Hospital ( Site 3603), Taipei
- Ukraine (4):
  - Municipal Enterprise "Bukovinian сlinical oncology сenter" ( Site 2504), Chernivtsi, Chernivetska Oblast
  - ME RIVNE REGIONAL ANTITUMOR CENTER ( Site 2517), Rivne, Rivne Oblast
  - Shalimov Institute of Surgery and Transplantation Oncology department ( Site 2512), Kyiv
  - Universal Clinic Oberig ( Site 2506), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/